CLINICAL TRIAL: NCT03533062
Title: Trigonal-sparing Versus Trigonal-involved Intravesical Botulinumtoxin A Injection in Refractory Idiopathic Detrusor Overactivity.
Brief Title: Trigonal vs Non Trigonal Botox Injection in OAB.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abdelbaset, principal investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OAB Botox injection
Record Dates: First submitted 2018-04-29; First posted 2018-05-22 (Actual); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Urologic Diseases; Overactive Bladder Syndrome; Quality of Life; Anticholinergic Syndrome
Keywords: OAB , Botox , anticholinergics , quality of life
MeSH Terms: conditions — Urologic Diseases; Anticholinergic Syndrome | interventions — Botulinum Toxins, Type A; Cholinergic Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- trigonal sparing botox injection (Active Comparator): Using a 7 gauge needle injection were allocated uniformly and evenly throughout the designed area excluding trigone in other arm Dilution of BOTOX vial (100 u) in 10 ml normal saline (10 u/ml) and injected in 20 sites (0.5ml /site).•then after 6 months postoperative anticholinergics administration .
  Interventions: Drug: botulinum toxin A
- trigonal involved (Active Comparator): Using a 7 gauge needle injection were allocated uniformly and evenly throughout the designed area including the trigone .Dilution of BOTOX vial (100 u) in 10 ml normal saline (10 u/ml) and injected in 20 sites (0.5ml /site).then after 6 months postoperative anticholinergics administration .
  Interventions: Drug: botulinum toxin A

INTERVENTIONS:
Drug: botulinum toxin A — botox A injection trigonal or trigonal sparing with trial of anticholinergics 6 months post operative for 3 months
  Other Names: anticholinergics

SUMMARY:
The investigators attend to conduct a prospective randomized study to assess safety and efficacy of trigonal-involved vs. trigonal-sparing botox injection technique, quality of life measurement and post-injection anticholinergics use efficacy.

Assessing safety by identification of side effects like constipation, urine retention....etc.

efficacy is measured using Over Active Bladder Symptoms Score(OABSS) and urodynamics measures after 6 months follow up.

DETAILED DESCRIPTION:
Overactive bladder (OAB) is a condition characterized by the presence of urinary urgency, typically joined by frequency and nocturia, with or without urgency urinary incontinence [UUI], in the absence of urinary tract infection (UTI) or other clear pathology.

Frequency is the most commonly reported symptom coming to 85% while 54% complained of urgency and 36% urgency incontinence.

OAB has usually resulted from detrusor over activities. The basic cause could be a neurological disorder (neurogenic type) such as spinal cord injuries, multiple sclerosis. In some cases, no obvious cause could be identified (idiopathic type).

OAB is a prevalent, chronic symptom complex that can impair quality of life (QOL). The prevalence of OAB in the general population was evaluated at 11.8% in a population-based survey conducted across five European countries. Epidemiological studies from North America have reported prevalence of OAB in women of 16.9% and the prevalence increases with age rising to 30.9% in those beyond 65 years.

Treatment objectives are to reduce the occurrence of bothersome symptoms. Several treatment choices are available for OAB including bladder and behavioral training, pharmacologic treatment, and surgical treatment.

Antimuscarinics are well established as pharmacotherapy for reducing OAB symptoms and enhancing QOL.Although, their use is limited in some patients by insufficient response to treatment "refractory OAB", or intolerable side effects , for example , dry mouth , blurred vision , constipation and cognitive impairment.

More recently, a European and Australian trial including about 2000 patients assessed mirabegron (β-3 agonist) (50 mg and 100 mg) in comparison to tolterodine (4 mg ER preparation) and placebo. There was a significant reduction in the number of voids over a 24-hours period, and incontinence episodes, vs. placebo at 12 weeks, at 1.93 vs. 1.34 (P < 0.05) and 1.57 vs. 1.17 (P < 0.05), respectively.

After a trial of pharmacotherapy, if the patient has not had satisfactory improvement in symptoms, intra-vesicle injection of Botox (BTX) can be offered as the following step.

Botulinum toxin (BTX) is a neurotoxin, it contains a heavy chain that binds to the presynaptic terminal of the neuromuscular junction , and this then acts by inhibiting the release of acetylcholine from the presynaptic vesicles at the axon terminal of the motor end plate , that then results in the muscle that is innervated becoming ﬂaccidly paralyzed. BTX is available in different preparations. The current commercially utilized type is BTX type A.

Now, there is cumulative data supporting use of BTX in cases of refractory Detrusor overactivity (DO).

Intradetrusal injection of BTX is followed by a significant improvements in the number of voiding episodes over 24 hours, incontinence episodes, urodynamic variables and quality of life scores. There is a decrease in episodes of urgency and incontinence by 80% and 60%, respectively. The efficacy peaks at 4 weeks, with the effect lasting typically up to 9 months.

Some essential issues for further investigations are the injection site, volume and number of injections. In terms of dosage, there are no firm recommendations, but in practice the advice was for a lower starting dose of 100 units of BTX-A, based on the currently available research. The disadvantage with higher dosing is the reduction in detrusor voiding pressures and an increased risk of voiding problems, while at the same time there is no increased efficacy.

The current AUA and EUA guidelines recommend trigonal sparing technique. During the injection process the trigone is typically spared because of the theoretical risk of de novo VUR from inhibition of the peritrigonal anti-reflux mechanism.

Moreover, trigonal area is rich in sensory fibers, therefore trigonal injection may enhance sensory component of urgency.

ELIGIBILITY:
Inclusion Criteria:

* Patients with idiopathic OAB refractory to treatment with antimuscarinics for 2 months or intolerable side effects of antimuscrinics

Exclusion Criteria:

* Patients who have any of the following were excluded:

  * Age less than 18 year old.
  * Neurogenic detrusor overactivity.
  * Evidence of obstructed flow in absence of prolapse.
  * Mixed urinary incontinence
  * Associated urethral pathology, e.g. Urethral diverticulum
  * Associated bladder pathology e.g. Fistula.
  * Active urinary tract infection as evidenced by positive urine culture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06-14 (Actual); Primary Completion 2016-10-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
efficacy of Botox injections of the bladder treating OAB using Over active bladder Symptoms score (OABSS).OABSS total score is 15.more score means more symptoms.it is divided into:1-5 &6-10&11-15 means mild &moderate&sever symptoms respectively. | 3 months
  Over active bladder symptoms score (OABSS).

SECONDARY OUTCOMES:
efficacy of anticholinergics post botox injection using Over active bladder symptoms score (OABSS). | 3 months
  Over active bladder symptoms score (OABSS).OABSS total score is 15.more score means more symptoms.it is divided into:1-5 &6-10&11-15 means mild &moderate&sever symptoms respectively.
quality of life assessment of patients with anticholinergics alone vs patients with botox injections vs combined therapy. | 3 months
  I-QOL Questionnaire
Arabic validation of overactive bladder symptoms score | 3 months
  To validate and translate English form to Arabic version of the over active bladder symptoms score (OABSS)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Shoma, MD, Study Chair — Urology and Nephrology Cente. Mansourah, Aldakahlia, Egypt, 35516

REFERENCES:
- [Derived] Elbaset MA, Hashem A, Taha DE, Zahran MH, El-Hefnawy AS. Validation of the Arabic linguistic version of the Overactive Bladder Symptoms Score questionnaire. Arab J Urol. 2019 Jun 12;17(4):265-269. doi: 10.1080/2090598X.2019.1627061. eCollection 2019. PMID 31723443